CLINICAL TRIAL: NCT00120315
Title: Proton Pump Inhibitor Treatment Stop: Discontinuation of Acid-suppressive Medication Among Long-term Users in a Primary Health Care Setting
Brief Title: Proton Pump Inhibitor Treatment Stop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Research Unit of General Practice, Odense (Other); University of Southern Denmark (Other); The Danish Medical Research Council (Other); Apotekerfonden af 1991 (Other); AstraZeneca (Industry); Danish College of General Practitioners (Other)
Responsible Party: Ove B. Schaffalitzky de Muckadell, prof., Odense University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2612-2176; MPU 16-2003; D9612L00060; 02.04; VF 20020212
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Dyspepsia
Keywords: dyspepsia; discontinuation; Primary health care; Helicobacter pylori; Proton Pump Inhibitor; Histamine-2-receptor-antagonist
MeSH Terms: conditions — Dyspepsia | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- esomeprazole (No Intervention): Long-term users continue antisecretory medication
  Interventions: Drug: esomeprazole; Procedure: Helicobacter pylori c-13 breath test
- placebo drug (Placebo Comparator): Long-term users are treated with placebo
  Interventions: Drug: esomeprazole; Procedure: Helicobacter pylori c-13 breath test

INTERVENTIONS:
Drug: esomeprazole — esomeprazole, original Nexium, 40 mg pills Up to once a day
Procedure: Helicobacter pylori c-13 breath test — Breath test done at entry to find Helicobacter pylori

SUMMARY:
The purpose of this study is to determine how many chronic users of antisecretory medication can stop after a test for a bacteria associated with peptic ulcer disease.

This is evaluated in a discontinuation trial.

DETAILED DESCRIPTION:
Background:

Testing patients with a Helicobacter pylori (Hp) 13C-urea breath test and treatment with eradication of Hp if positive - test-and-eradicate - have proven as effective and safe as prompt endoscopy for management of dyspeptic patients in a primary health care setting. However, empirical treatment with an ulcer-healing drug is often used in dyspeptic patients, as reflected in a growing proportion of long-term users without known ulcer or gastro-oesophageal reflux disease (GORD). This group of patients contributed to 59% of the total use of acid-suppressive medication in the County of Funen in Denmark in 1997.

Aim/purpose:

It is our aim to examine the need for continued medication with prescribed, acid-suppressive drugs in primary health care.

Our secondary objective is to investigate the profile of symptoms, quality of life, Hp-status, consumption of drugs and use of health care services in the same context.

Methods:

To conduct a randomised, placebo-controlled, blinded, clinical discontinuation trial, 500 long-term users of acid-suppressive drugs are identified by general practitioners. Long-term use is defined as treatment for more than 2x28 days during a 6-month period. The patients are included with a 13C-urea Hp-breath test and randomised for treatment with PPI or placebo. Hp-positive patients are treated with an Hp-eradication treatment. The patients are followed for 1 year; the primary outcome is the need for open treatment with acid-suppressive medication due to failing symptom relief despite treatment with the randomised project medication. The patients are to fill in a symptom and medication diary every month for periods of 1 week. Questionnaires are to be given to the patients 3 times during the follow-up period. Medication diaries as well as questionnaires have proven useful in similar studies. The main outcome is analysed using Kaplan-Meier survival estimates analysis.

ELIGIBILITY:
Inclusion Criteria:

* Use of antisecretory medication for more than 2 months during the last 6 months

Exclusion Criteria:

* Malignity or severe, competing medical or psychiatric disease
* Esophagitis (proven by endoscopy)
* Prior complication to peptic ulcer disease
* Alarm symptoms
* Pregnancy or lactation
* Allergy towards esomeprazole
* Planned hospitalisation during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Failure of patient perceived symptom control despite treatment with project medication | 12 months

SECONDARY OUTCOMES:
Gastrointestinal symptoms | 12 months
Quality of life | 12 months
GPs and patients satisfaction | 12 months
Helicobacter pylori status | At enrolement
Resource consumption | 12 months
Days without symptoms | 12 months
Use of otc-medication | 12 months
Sick-leave days | 12 months
Number of visits to primary and secondary healthcare system | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ove B Schaffalitzky de Muckadell, Professor, Study Director — Odense University Hospital
Locations (1):
- Department of Medical Gastroenterology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Zwisler JE, Jarbol DE, Lassen AT, Kragstrup J, Thorsgaard N, Schaffalitzky de Muckadell OB. Placebo-Controlled Discontinuation of Long-Term Acid-Suppressant Therapy: A Randomised Trial in General Practice. Int J Family Med. 2015;2015:175436. doi: 10.1155/2015/175436. Epub 2015 Jul 12. PMID 26246908